CLINICAL TRIAL: NCT06732934
Title: The Effect of Basic Body Awareness Therapy and Aerobic Exercise Approaches on Telomere Length in Young Individuals
Brief Title: Body Awareness and Aerobic Exercise: Telomere Impact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Mert Usta, RA, Research Asistant, Suleyman Demirel University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BBAT
Record Dates: First submitted 2024-11-21; First posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Exercise
Keywords: aerobic exercise; basic body awareness therapy; telomere lenght
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: In this study, a parallel group design is used, where participants are randomly assigned to one of three independent groups:
  Basic Body Awareness Therapy Group Aerobic Exercise Group Control Group Each group receives a different intervention (body awareness therapy, aerobic exercise, or no intervention for the control group) and is observed over the study period. The study aims to compare the effects of body awareness therapy and aerobic exercise on telomere length in young individuals. The control group serves to assess the natural variation in telomere length without any intervention. This design allows for a clear comparison of the outcomes between the different groups, ensuring that any observed effects can be attributed to the specific intervention each group received.
  In summary, each group follows its own intervention pathway independently, and the results from each group are analyzed to understand the impact on telomere length.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Basic Body Awareness Therapy Group (Experimental): Participants will engage in 12 weeks of Basic Body Awareness Therapy (BBAT) three times a week. The exercises will include body scanning, stretching, strength accumulation, sound resonance, and midline orientation, supervised by an experienced physiotherapist. Each session lasts 40 minutes, with 5 minutes of meditation and a group feedback session after every exercise. The group will consist of a maximum of 10 participants.
  Interventions: Other: exercise (Basic Body Awareness Therapy
- Aerobic Exercise Group (Experimental): Participants will undergo aerobic exercise on a treadmill, following ACSM guidelines. Exercise duration will start at 30 minutes in the first week and gradually increase to 45 minutes by the 12th week. The exercise intensity will be monitored using the target heart rate method (64-77% HRmax) and will be supervised by a physician. Heart rate monitoring will be done during the exercises, and participants will be asked to maintain their usual diet.
  Interventions: Other: exercise (aerobic exercise)
- Control Group (No Intervention): No intervention or recommendations will be provided to the control group.

INTERVENTIONS:
Other: exercise (Basic Body Awareness Therapy — Body Awareness Therapy is a patient-centered physiotherapy approach that also includes mental health, focusing on movement awareness training. This therapy primarily consists of exercises aimed at improving postural disorders, balance, and muscle tension. It aims to help individuals experience and accept bodily responses while increasing coping strategies.
  The therapy includes body scanning, integration of sound and movement, stretching exercises, and exercises focusing on body alignment and midline orientation.
  Floor exercises: body scanning, stretching, strength accumulation, sound resonance.
  Seated exercises: body alignment, trunk rotation, head and neck movements. Standing exercises: support surface perception, midline elevation and lowering, bilateral arm movements, rotation, one-legged balance, voice exercises, and group movements.
  Arms: Basic Body Awareness Therapy Group
Other: exercise (aerobic exercise) — The continuous exercise protocol specified by the American College of Sports Medicine (ACSM) will be applied under supervision on a treadmill. The exercise duration will follow ACSM recommendations, starting at 30 minutes in the first week and increasing to 45 minutes by the 12th week.
  Exercise intensity will be assessed using the target heart rate method (220 - age). The intensity of aerobic exercise will be set at a moderate level (64-77% HRmax), according to ACSM guidelines.
  During exercise, heart rate will be monitored through a heart rate monitoring device. A 5-minute warm-up and a 5-minute cool-down exercise will be performed before and after each session, with an intensity of 50-60% of the maximum heart rate.
  Arms: Aerobic Exercise Group

SUMMARY:
Telomeres shorten with each replication cycle throughout cellular lifespan. While it is known that telomere length is age-dependent, numerous factors influencing telomere length have been identified. One such factor is the perception of stress created by the individual and their environment. It has been suggested that stress and depression can alter telomere structure by increasing pro-inflammatory cytokines. The aim of this study is to preserve healthy telomere structure by controlling stress levels. In this context, Basic Body Awareness Therapy (BBAT) exercises, known to be more effective than standard exercise approaches in reducing stress and depression, will be used as an alternative. There are no studies in the literature examining the effects of BBAT on epigenetic mechanisms. This study aims to contribute to the existing literature by comparing BBAT with aerobic exercise, which is recognized as one of the most effective exercise approaches for preserving telomere structure. Furthermore, the hypothesis that telomere length changes, observed over a long period in previous studies, can be achieved in a shorter time through BBAT-an approach known to be more effective in stress management based on mind-body principles-represents one of the unique aspects of this research. The study aims to provide valuable insights into identifying the most effective exercise approaches for influencing telomere length changes

DETAILED DESCRIPTION:
Telomeres are specialized regions located at the ends of chromosomes that allow chromosomal replication. In most human somatic cells, telomeres naturally shorten with each successive cell division. While telomere shortening is known to be age-dependent, numerous internal and external factors that influence telomere length have been identified. Genetic factors, such as DNA methylation, contribute to internal factors, while external factors include lifestyle practices, such as diet and exercise, that induce epigenetic changes and facilitate genomic regulation.

High levels of stress are associated with shorter telomere length, as stressors can disrupt telomere structure through a series of chemical reactions. Consequently, lifestyle changes or interventions that reduce stress levels have been widely explored. The common focus of these studies involves factors that protect telomeres and regulate telomerase activity. This study aims to preserve healthy telomere structure by controlling stress levels.

Stressors change with age, and emotional distress, interpersonal rejection, financial concerns, and feelings of social exclusion in younger individuals are known to elevate stress levels. Additionally, younger individuals' psychological responses to stress tend to be more intense. This can directly affect emotional responses, behavioral coping, emotional regulation, and rumination. Since the core of stress lies in human perception and evaluation of experiences, how an individual interprets, assesses, and responds to these experiences becomes critical in stress management. Therefore, this study adopts an approach that addresses these factors for stress management.

Studies on telomere length changes associated with physical activity and exercise suggest that more active individuals tend to have longer telomeres. However, moderate activity levels have been associated with longer telomeres compared to inactive or excessively active individuals. Woo et al. did not find a difference in telomere length between inactive and active individuals, but their study focused on elderly populations.

Research on stress levels and telomere length has shown that individuals with lower stress levels tend to have longer telomeres. Likewise, meditation practices are reported to regulate psychological mediators by enhancing telomerase activity in immune cells. Blackburn's study found that chronic psychological stress, its perception, and high oxidative stress were associated with shorter telomeres, lower telomerase activity, and cell aging in healthy peripheral mononuclear blood cells.

Studies comparing exercise interventions have indicated that resistance training does not alter telomere length. Since endurance and resistance training did not produce changes in telomere length, alternative exercise approaches were proposed. While some studies suggest that short-term aerobic exercise does not change telomere length, aerobic exercise, both short and long term, is recognized as a significant exercise type that contributes to telomere elongation. Mind-body interventions to preserve telomere structure have been limited, with most research focusing on meditation and yoga. However, promising studies on meditation have been conducted, with one study showing telomere length increase after 12 weeks of meditation training.

Although telomere structure is primarily influenced by age and genetics, factors such as smoking, alcohol consumption, lifestyle changes, diet, and chronic inflammatory processes can also affect telomere structure. Based on the existing literature, this study aims to investigate the effects of TBFT (Basic Body Awareness Therapy) and aerobic exercise on high-stress individuals, while controlling for secondary factors as much as possible, to determine the effectiveness of these exercises.

This study aims to track changes in telomere length in high-stress young individuals using standard aerobic exercise and basic body awareness exercises (BBAT).

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 18-30,
* Not be obese (BMI < 25 kg/m²),
* Not have a history of regular exercise or long-term exercise participation,
* Not have a history of smoking or alcohol use,
* Not have received hormone replacement therapy,
* Not be using antioxidant or multivitamin supplements,
* Not have a diagnosed acute or chronic inflammatory disease or any rheumatic condition,
* Be willing to participate in the study voluntarily

Exclusion Criteria:

* Having been diagnosed with a severe psychiatric disorder or using psychiatric medication,
* Having communication barriers,
* Having a history of smoking or alcohol use,
* Having a history of regular exercise,
* Having variable general nutrition habits,
* Having any other diseases related to the circulatory system, orthopedic, neurological, cardiac, and respiratory functions, such as diabetes, cholesterol, or heart failure,
* Being enrolled in another exercise program during the 12-week period within the assigned exercise group.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Telomere Length Measurement | 3 months
  Blood samples will be collected by Dr. Faculty Member Halil ÖZBAŞ at the SDU Research Application Hospital's medical genetics laboratory and will be properly stored. DNA will be isolated from a 2cc peripheral venous blood sample collected in an EDTA tube using a DNA isolation kit and an appropriate protocol. After measuring the DNA's purity and concentration, suitable DNA samples will be used for telomere copy number measurement with a Real-Time PCR method using a telomere copy number measurement kit.
  Telomere length will be assessed twice, once before and once after the 12-week exercise program.
Perceived Stress Scale | 3 months
  The scale consists of 14 items in total. It is designed to measure the degree to which certain situations in an individual's life are perceived as stressful. Each item on the scale is rated on a 5-point Likert-type scale ranging from "Never (0)" to "Very Often (4)." Seven of the items that contain positive expressions are reverse scored. The scores of the PSS-14 range from 0 to 56. A high score indicates a high level of stress perception. The PSS consists of two subscales: inadequate self-efficacy and stress/discomfort perception. A score between 11-26 indicates a low level of stress, between 27-41 indicates a moderate level of stress, and between 42-56 indicates a high level of stress
Beck Depression Inventory | 3 months
  Developed by Beck et al., the Turkish validity and reliability of the scale has been established. It consists of 21 questions, and the scores for each response, ranging from 0 to 3, are summed to determine the overall score. The highest possible score is 63, and a higher score indicates a higher severity of depression.
Beck Anxiety Inventory | 3 months
  Developed by Beck et al. and adapted into Turkish, this scale consists of 21 questions. Each question is rated on a scale from 0 to 3, and the total score is used to assess the severity of anxiety symptoms. The total score ranges from 0 to 63
Body Awareness Questionnaire | 3 months
  The body awareness questionnare is a valid and reliable scale in Turkish used to measure body awareness. It evaluates body awareness in four distinct subdimensions: the ability to identify changes in the body or changes in response to specific stimuli, the ability to predict responses to certain stimuli, awareness of sleep and wake cycles and sleep duration, and the ability to sense illness before it manifests. The questionnaire consists of 18 questions, which aim to measure changes across these four subdimensions. For each question, individuals are asked to select the most appropriate answer from 8 options, ranging from 0 (this statement is not true for me) to 7 (this statement is completely true for me). The result is expressed as the total score from the items, with higher scores indicating better body awareness.
Pittsburgh Sleep Quality Index | 3 months
  The Pittsburgh Sleep Quality Index (PSQI) will be used to assess patients' sleep quality, a valid and reliable method in Turkish. The PSQI consists of 24 questions directed to the patient to define sleep quality as good or poor. Of these questions, 19 are self-assessment items answered by the patient, while the remaining 5 are answered by the patient's spouse or roommate. The PSQI score is calculated based on the total score, excluding the 5 questions answered by others. The 19 self-assessment questions evaluate various aspects of sleep quality, including sleep duration, sleep onset delay, and the frequency and severity of specific sleep-related issues.
Ruminasyon Scale | 3 months
  The Ruminasyon Scale, developed by Nolen-Hoeksema and Morrow, consists of 10 items. It is a 4-point Likert scale (never, sometimes, often, always). The scale has two subdimensions: deep thinking and obsessive thinking. The maximum score that can be obtained from the scale is 40, and the minimum score is 10. A higher score indicates more rumination. The Turkish adaptation and validity-reliability study of the Ruminasyon Scale was conducted by Erdur-Baker and Bugay, and it was examined for high school and university students
SF-12 Quality of Life Scale | 3 months
  The Turkish validated and reliable version of the Short Form-12 (SF-12) Health Survey will be used to assess individuals' quality of life. The SF-12 is a shorter version of the original 36-item Health Survey, containing 12 selected items. The scale evaluates eight subdimensions: physical functioning, role limitations due to physical health, social functioning, pain, mental health, role limitations due to emotional problems, vitality, and general health perception. These subdimensions are combined into two main domains: physical health and mental health. Patients rate their experiences over the past month on a scale of 1 to 3 for some items and 1 to 5 for others. Scores for the eight subdimensions and two main domains are calculated separately and expressed as percentages, with a score of 100% indicating optimal quality of life. Responses will be scored using an open-access online calculator available at orthotoolkit.com/sf-12.

CONTACTS AND LOCATIONS:
Overall Officials: Mert Usta, RA, Principal Investigator — https://w3.sdu.edu.tr/personel/06713
Locations (1):
- Süleyman Demirel University, Isparta, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data is intended to be used solely within the scope of the specified research questions, and sharing it beyond this scope is deemed inappropriate.

REFERENCES:
- [Background] Tosato M, Zamboni V, Ferrini A, Cesari M. The aging process and potential interventions to extend life expectancy. Clin Interv Aging. 2007;2(3):401-12. PMID 18044191
- [Background] Kanherkar RR, Stair SE, Bhatia-Dey N, Mills PJ, Chopra D, Csoka AB. Epigenetic Mechanisms of Integrative Medicine. Evid Based Complement Alternat Med. 2017;2017:4365429. doi: 10.1155/2017/4365429. Epub 2017 Feb 21. PMID 28316635
- [Background] Jacobs TL, Epel ES, Lin J, Blackburn EH, Wolkowitz OM, Bridwell DA, Zanesco AP, Aichele SR, Sahdra BK, MacLean KA, King BG, Shaver PR, Rosenberg EL, Ferrer E, Wallace BA, Saron CD. Intensive meditation training, immune cell telomerase activity, and psychological mediators. Psychoneuroendocrinology. 2011 Jun;36(5):664-81. doi: 10.1016/j.psyneuen.2010.09.010. Epub 2010 Oct 29. PMID 21035949
- [Background] Scarabino D, Peconi M, Broggio E, Gambina G, Maggi E, Armeli F, Mantuano E, Morello M, Corbo RM, Businaro R. Relationship between proinflammatory cytokines (Il-1beta, Il-18) and leukocyte telomere length in mild cognitive impairment and Alzheimer's disease. Exp Gerontol. 2020 Jul 15;136:110945. doi: 10.1016/j.exger.2020.110945. Epub 2020 Apr 11. PMID 32289486
- [Background] Cherkas LF, Hunkin JL, Kato BS, Richards JB, Gardner JP, Surdulescu GL, Kimura M, Lu X, Spector TD, Aviv A. The association between physical activity in leisure time and leukocyte telomere length. Arch Intern Med. 2008 Jan 28;168(2):154-8. doi: 10.1001/archinternmed.2007.39. PMID 18227361
- [Background] Ludlow AT, Zimmerman JB, Witkowski S, Hearn JW, Hatfield BD, Roth SM. Relationship between physical activity level, telomere length, and telomerase activity. Med Sci Sports Exerc. 2008 Oct;40(10):1764-71. doi: 10.1249/MSS.0b013e31817c92aa. PMID 18799986
- [Background] Woo J, Tang N, Leung J. No association between physical activity and telomere length in an elderly Chinese population 65 years and older. Arch Intern Med. 2008 Oct 27;168(19):2163-4. doi: 10.1001/archinte.168.19.2163. No abstract available. PMID 18955647
- [Background] Puterman E, Lin J, Blackburn E, O'Donovan A, Adler N, Epel E. The power of exercise: buffering the effect of chronic stress on telomere length. PLoS One. 2010 May 26;5(5):e10837. doi: 10.1371/journal.pone.0010837. PMID 20520771
- [Background] O'Donovan A, Tomiyama AJ, Lin J, Puterman E, Adler NE, Kemeny M, Wolkowitz OM, Blackburn EH, Epel ES. Stress appraisals and cellular aging: a key role for anticipatory threat in the relationship between psychological stress and telomere length. Brain Behav Immun. 2012 May;26(4):573-9. doi: 10.1016/j.bbi.2012.01.007. Epub 2012 Jan 24. PMID 22293459
- [Background] Werner CM, Hecksteden A, Morsch A, Zundler J, Wegmann M, Kratzsch J, Thiery J, Hohl M, Bittenbring JT, Neumann F, Bohm M, Meyer T, Laufs U. Differential effects of endurance, interval, and resistance training on telomerase activity and telomere length in a randomized, controlled study. Eur Heart J. 2019 Jan 1;40(1):34-46. doi: 10.1093/eurheartj/ehy585. PMID 30496493
- [Background] Ribeiro VB, Pedroso DCC, Kogure GS, Lopes IP, Santana BA, Dutra de Souza HC, Ferriani RA, Calado RT, Furtado CLM, Reis RMD. Short-Term Aerobic Exercise Did Not Change Telomere Length While It Reduced Testosterone Levels and Obesity Indexes in PCOS: A Randomized Controlled Clinical Trial Study. Int J Environ Res Public Health. 2021 Oct 27;18(21):11274. doi: 10.3390/ijerph182111274. PMID 34769797
- [Background] Innes KE, Selfe TK, Brundage K, Montgomery C, Wen S, Kandati S, Bowles H, Khalsa DS, Huysmans Z. Effects of Meditation and Music-Listening on Blood Biomarkers of Cellular Aging and Alzheimer's Disease in Adults with Subjective Cognitive Decline: An Exploratory Randomized Clinical Trial. J Alzheimers Dis. 2018;66(3):947-970. doi: 10.3233/JAD-180164. PMID 30320574
- [Background] Song S, Lee E, Kim H. Does Exercise Affect Telomere Length? A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Medicina (Kaunas). 2022 Feb 5;58(2):242. doi: 10.3390/medicina58020242. PMID 35208566